CLINICAL TRIAL: NCT04732481
Title: Evaluation of Corrected Carotid Flow Time Variations During Passive Leg Lift to Predict Response to Filling
Acronym: CAROT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cornouaille (Other)
Responsible Party: Sponsor
Other Study IDs: QP-RIPH3-001
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Organ Failure, Multiple
MeSH Terms: conditions — Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- interventional group: passive leg lift test
  Interventions: Procedure: passive leg lift test
- control group: no intervention (SOC)

INTERVENTIONS:
Procedure: passive leg lift test — passive leg lift test
  Groups: interventional group

SUMMARY:
Patients hospitalized in intensive care often require intravenous administration of fluid in order to optimize the functioning of the heart and thus ensure perfusion of vital organs such as the kidneys, the brain or the digestive tract. However, it is necessary to find the right balance in fluid intake because it has been shown that excessive administration has a negative impact on patient survival, the length of their stay in intensive care or the duration of invasive mechanical ventilation.The passive leg lifting maneuver is regularly used to determine which patients should be infused with these large volumes (the patient's chest is placed in a horizontal position and the legs are elevated at 30 ° by tilting the bed for 2 minutes ). To be interpreted, this maneuver requires the presence of invasive devices (bloody arterial pressure catheter, PICCO monitor) or an operator experienced in cardiac ultrasound.Our study aims to evaluate an easy-to-use, non-invasive tool widely available in intensive care and emergency departments (carotid vascular doppler ultrasound) to assess the response to a passive leg lifting maneuver. . The measurements are taken before and after a passive leg lifting maneuver and then before and after a filling decided before inclusion by the doctor responsible for the patient.

ELIGIBILITY:
Inclusion Criteria:

* equipped with a PICCO2® continuous cardiac output monitoring device
* for which the practitioner in charge of the patient decides to administer a volume expansion

Exclusion Criteria:

* patients whose rhythm is non-sinus
* who have expressed their refusal to participate in the protocol
* contraindicated to passive leg lifting maneuvers (deep vein thrombosis, HTIC, BMI> 40 or> 14, spinal instability)
* pregnant women and patients clinically suspected of abdominal compartment syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: During their ICU admission for organ failure or multiple organ failure, patients frequently receive volume expansion to increase cardiac output.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
response to filling | 90sec
  Collection of the diagnosis of response to filling after volume expansion of 500mL of Isotonic Salted Serum and evaluation of the variation in TFCc during passive leg lifting between the two groups

SECONDARY OUTCOMES:
cut-off value for positivity of the test | 90sec
  The secondary objective of this work is to determine the best positivity threshold value of the test studied as well as its sensitivity and specificity for the chosen value.

CONTACTS AND LOCATIONS:
Locations (1):
- Ch Cornouaille, Quimper, Finistere, France